CLINICAL TRIAL: NCT06817603
Title: Comparison of Procedural Oxygen Mask vs. High-flow Nasal Cannula for Hypoxemia Prevention During Endoscopic Retrograde Cholangiopancreatography (ERCP): A Randomized Parallel-GroupTrial
Brief Title: Procedural Oxygen Mask vs. High-flow Nasal Cannula for Hypoxemia Prevention During ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Principal Investigator, Bedirhan Günel, Principal Investigator, Kocaeli City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KSH-ANREA-BG-05
Record Dates: First submitted 2025-01-31; First posted 2025-02-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Hypoxemia
Keywords: Hypoxemia; Endoscopic Retrograde Cholangiopancreatography; Airway Management
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (Active Comparator): Oxygen administered during the endoscopic retrograde cholangiopancreatography (ERCP) procedure will be delivered through a Procedural Oxygen Mask (POM® ELITE MF). The procedural oxygen mask is a device that covers both the mouth and nose to deliver oxygen to the patient. Its reservoir feature increases the concentration of delivered oxygen
  Interventions: Device: Procedural Oxygen Mask
- Group H (Active Comparator): During the Endoscopic Retrograde Cholangiopancreatography (ERCP) procedure, oxygen will be delivered through a High-Flow Nasal Cannula (HFNC) device. The high-flow nasal cannula is a device that provides humidified and heated oxygen to the patient via the nasal route. Its high flow rate increases the fraction of inspired oxygen (FiO₂), ensuring more effective oxygenation and reducing dead space ventilation.
  Interventions: Device: High-Flow Nasal Cannula

INTERVENTIONS:
Device: Procedural Oxygen Mask — Procedural Oxygen Mask will be used
  Arms: Group P
Device: High-Flow Nasal Cannula — High-Flow Nasal Cannula (HFNC) will be used.
  Arms: Group H

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is an imaging procedure that visualizes the drainage ducts of the pancreas, gallbladder, and liver through the use of a duodenoscope and contrast media. By endoscopically identifying the ampulla of Vater, the common bile duct is cannulated. ERCP is also frequently utilized for therapeutic interventions, such as endoscopic sphincterotomy, bile duct stone extraction, stent placement in malignant and benign biliary strictures, and biopsy collection, thus playing a critical role in both the diagnosis and treatment of pancreatobiliary disorders.

ERCP, being more invasive than routine upper endoscopies or colonoscopies, typically necessitates deeper levels of sedation. The procedure is performed in the prone, modified prone, or lateral decubitus position, which increases the risk of hypoxemia and hypoventilation due to upper airway obstruction. Furthermore, endoscopic instruments inserted through the oral cavity limit anesthesiologists' access to the patient's airway, thereby restricting ventilation support during gastrointestinal endoscopy. Ensuring airway stability during sedation is paramount for patient safety and procedural efficacy. Currently, a range of devices, including traditional nasal cannulas, high-flow oxygen masks, and procedural oxygen masks, are employed to provide oxygen support throughout the procedure.

The existing literature includes randomized controlled trials and systematic reviews aimed at preventing hypoxemia during ERCP. Through this study, investigators aim to make a novel contribution to the literature by assessing the effectiveness of a recently introduced procedural oxygen mask.

DETAILED DESCRIPTION:
This study aims to compare the efficacy of two oxygen delivery methods-High-Flow Nasal Cannula (HFNC) and Procedural Oxygen Mask (POM)-in preventing hypoxemia during Endoscopic Retrograde Cholangiopancreatography (ERCP). Designed as a randomized, parallel-group, prospective study, participants were assigned to two groups, Group H (HFNC) and Group P (POM), in a 1:1 ratio using computer-assisted random allocation. However, due to the visible differences between the oxygen delivery devices, neither healthcare providers nor patients could be blinded to the randomization.

The study was planned to include 134 patients (67 per group) with a 95% confidence level (1-α) and 90% test power (1-β). To account for an anticipated 10% dropout rate, the total sample size was set at 150 patients.

Throughout the ERCP procedure, all patients will be monitored using pulse oximetry, electrocardiography (ECG), and non-invasive blood pressure monitoring. Capnography will be applied in both groups, and necessary interventions will be carried out by anesthesia specialists if a patient's oxygen saturation falls below 90%. All interventions and events will be meticulously documented. Following the procedure, patients will be monitored in the post-anesthesia care unit (PACU), and those with a Modifiye Alderete score of 10 will be discharged.

The FiO2 will be maintained constant throughout the procedure. Patients will initially receive midazolam at a dose of 0.02 mg/kg, followed by 0.5 mg/kg of ketamine. To ensure adequate sedation, propofol will be administered as an initial bolus dose of 0.5-1.0 mg/kg, with additional boluses of 0.25-0.5 mg/kg every 1-3 minutes as needed to maintain the target sedation level.

The target sedation depth will be 3-4 on the Ramsay Sedation Scale (RSS), and this level will be maintained throughout the procedure. Upon completion, patients will be awakened using verbal and tactile stimuli. Once their RSS reaches 2, they will be transferred to the Post-Anesthesia Care Unit (PACU). Patients will be discharged from the PACU upon achieving a Modified Aldrete Score (MAS) of 10.

Vital signs, procedure durations, and dosages of medications used for each patient will be meticulously recorded. All anesthesia-related decisions during the procedure will be made by the supervising anesthesia specialist.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years
* American Society of Anesthesiologists (ASA) classification of 1-2-3
* Patients scheduled for ERCP at Kocaeli City Hospital Endoscopy Unit

Exclusion Criteria:

* Refused to participate in the study
* Had an allergy to ketamine, propofol, or midazolam
* Had a BMI >30 kg/m²
* Were pregnant or in the postpartum period
* Had a STOP-BANG score ≥3
* Had a history of intubation within the past 3 months
* Had a history of lower respiratory tract infection within the past 3 months
* Had a history of intensive care unit (ICU) admission within the past 3 months
* Had a tracheostomy or a history of tracheostomy placement
* Were oxygen-dependent
* Had lung cancer or a history of lung surgery
* Had asthma, COPD, or interstitial lung disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
incidence of hypoxemia | Continuous SpO2 monitoring will be performed throughout the ERCP procedure
  The incidence of hypoxemia during sedation (defined as SpO2 < 90%). SpO₂ will be continuously measured using a pulse oximeter (GE Healthcare) to monitor and record oxygen saturation levels throughout sedation.

SECONDARY OUTCOMES:
Number of hypoxemia episodes | Continuous SpO2 monitoring will be performed throughout the ERCP procedure
  An episode was recorded when SpO2 dropped below 90% after reaching a level of SpO2 ≥ 90% for 30 seconds. SpO₂ will be continuously measured using a pulse oximeter (GE Healthcare) to monitor and record oxygen saturation levels throughout sedation.
Duration of hypoxemia | Continuous SpO2 monitoring will be performed throughout the ERCP procedure
  Defined as the time taken to reach SpO2 ≥ 90%. SpO₂ will be continuously measured using a pulse oximeter (GE Healthcare) to monitor and record oxygen saturation levels throughout sedation.
Continuous SpO2 monitoring will be performed throughout the ERCP procedure | Continuous SpO2 monitoring will be performed throughout the ERCP procedure
  Minimum SpO2 value observed during the procedure. SpO₂ will be continuously measured using a pulse oximeter (GE Healthcare) to monitor and record oxygen saturation levels throughout sedation.
Frequency of Chin Lift Maneuver | Interventions related to airway management causing interruptions during the procedure
  This outcome measure will assess the frequency of the chin lift maneuver performed during the procedure due to hypoxemia
Frequency of Jaw Thrust Maneuver | Interventions related to airway management causing interruptions during the procedure
  This outcome measure will assess the frequency of the Jaw Thrust maneuver performed during the procedure due to hypoxemia
Frequency of Mask Ventilation | Interventions related to airway management causing interruptions during the procedure
  This outcome measure will assess the frequency of the Mask Ventilation performed during the procedure due to hypoxemia
Frequency of Need for Aspiration | Interventions related to airway management causing interruptions during the procedure
  This outcome measure will assess the frequency of need for aspiration performed during the procedure due to hypoxemia
Frequency of High-Flow Nasal Cannula or Procedural Oxygen Mask (POM) Repositioning | Interventions related to airway management causing interruptions during the procedure
  This outcome measure will assess the frequency of Frequency of High-Flow Nasal Cannula or Procedural Oxygen Mask (POM) Repositioning during the procedure due to hypoxemia
Other potential complications | during the procedure
  Other potential complications that may arise during the procedure (hypotension, hypertension, bradycardia, tachycardia, movements that hinder the procedure) (Hypotension is defined as a decrease in the patient's baseline systolic blood pressure of more than 20% or a drop below 90 mm Hg. Hypertension is defined as an increase in the patient's baseline systolic blood pressure of more than 20%. A heart rate below 60 beats per minute is considered bradycardia, while a rate above 100 beats per minute is classified as tachycardia)
Gastroenterologist satisfaction | with data reported immediately following the completion of the procedure
  a 10-point scoring system was used, where 0 indicates "unmanageable, numerous interruptions or terminated procedure," and 10 indicates "excellent sedation, no interruptions"
Patient satisfaction related to anesthesia | Data will be recorded until discharge from the PACU, which is expected to occur within up to 2 hours after the procedure
  Patient satisfaction related to anesthesia was assessed and recorded before discharge (a scale from 0 to 10 was used, where 0 means "very poor, I would never undergo this procedure again," and 10 means "excellent, I would undergo this procedure again in the same manner
Dry mouth/nose/throat: | Data will be recorded until discharge from the PACU, which is expected to occur within up to 2 hours after the procedure
  Before discharge, patients in the Post-Anesthesia Care Unit (PACU) will be assessed for dry mouth, nose, and throat

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli City Hospital, Kocaeli, İ̇zmi̇t, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data will not be shared

REFERENCES:
- [Background] Nay MA, Fromont L, Eugene A, Marcueyz JL, Mfam WS, Baert O, Remerand F, Ravry C, Auvet A, Boulain T. High-flow nasal oxygenation or standard oxygenation for gastrointestinal endoscopy with sedation in patients at risk of hypoxaemia: a multicentre randomised controlled trial (ODEPHI trial). Br J Anaesth. 2021 Jul;127(1):133-142. doi: 10.1016/j.bja.2021.03.020. Epub 2021 Apr 28. PMID 33933271